CLINICAL TRIAL: NCT02842073
Title: Assessing Changes in the Brain Melanocortin System and Sensory Processing in Response to Alcohol to Advance Our Understanding of the Pathophysiology and Psychopharmacology of Binge Drinking
Brief Title: An Open Label Trial of Bupropion and Naltrexone for Binge Drinking
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-1370; TTSA018P1 (Other: NCTraCS)
Record Dates: First submitted 2016-06-15; First posted 2016-07-22 (Estimated); Results first posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-06

CONDITIONS: Binge Drinking
MeSH Terms: conditions — Binge Drinking | interventions — Naltrexone; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Naltrexone and Buproprion (Experimental): Investigators will use standard clinical doses of bupropion-XL 300 mg/d (lower seizure risk) and naltrexone 50 mg/d dispensed by the UNC Investigational Drug Services. Bupropion XL will be initiated at 150 mg/d on Days 1-4 and increased to 300 mg/d for Days 5-84. Naltrexone will be initiated at 25 mg/d from Days 7-9 and then go to 50 mg/d for Days 10-84.
  Interventions: Drug: Naltrexone; Drug: Bupropion

INTERVENTIONS:
Drug: Naltrexone — Standard clinical doses of naltrexone 50 mg/d dispensed by the UNC Investigational Drug Services. Naltrexone will be initiated at 25 mg/d from Days 7-9 and then go to 50 mg/d for Days 10-84.
Drug: Bupropion — Standard clinical doses of bupropion-XL 300 mg/d (lower seizure risk) dispensed by the UNC Investigational Drug Services. Bupropion XL will be initiated at 150 mg/d on Days 1-4 and increased to 300 mg/d for Days 5-84.

SUMMARY:
This is an open-label Phase IIa pilot study of the tolerability and effects on binge drinking of bupropion and naltrexone for binge drinkers.

DETAILED DESCRIPTION:
This is an open-label Phase IIa pilot study of the tolerability and effects on binge drinking of bupropion and naltrexone for binge drinkers.

Participants: Investigators will recruit 12 men or women ages 21-34 years who exhibit a minimum of 5/3 (men/women) or more binge drinking episodes per month over the past three months. A binge drinking episode is defined as the consumption of 5/4 (men/women) standard drinks (~12 gms ethanol) in about a two hour period. Subjects may meet DSM-V criteria for mild or moderate alcohol use disorder. Subjects with overt physical dependence on alcohol, significant medical problems including seizures or bulimia, other substance use disorder except for occasional marijuana (based on toxicology screen) or significant psychiatric illness will be excluded.

Procedures (methods): As a first step in human trials investigators will give open label bupropion + naltrexone to active binge drinking subjects. The primary goal here is to assess tolerability and acceptability though changes in binge drinking and subjective sense of "effect" will be gathered as well. Investigators will also test cortical adaptation to binge drinking by completing tactile sensory testing and comparing the results to controls and individuals with overt physical dependence on alcohol. Investigators will recruit subjects using the e-mail listserve for UNC students, faculty and staff.

Investigators will use standard clinical doses of bupropion-XL 300 mg/d (lower seizure risk) and naltrexone 50 mg/d dispensed by the UNC Investigational Drug Services. Bupropion XL will be initiated at 150 mg/d on Days 1-4 and increased to 300 mg/d for Days 5-84. Naltrexone will be initiated at 25 mg/d from Days 7-9 and then go to 50 mg/d for Days 10-84. Subjects will be seen at screening and then at Weeks 0, 1, 3, 5, 8 and 12. Subjects will be breathalyzed and receive Medical Management counseling to encourage compliance and progress towards drinking goals. Investigators will use the Time Line Follow-Back approach to assess alcohol consumption history modified to include time taken to consume alcohol and define a binge. They will also measure craving for alcohol and will assess tolerability by probing for adverse effects. Key outcomes of interest include tolerability and acceptability, drinking behavior including frequency and intensity of binge drinking, and craving for alcohol. Because this is an open-label trial without a placebo comparison group no formal statistics will be completed and efficacy will not be assessed. Instead, this pilot study will inform investigators about the recruitment of binge drinkers, the tolerability and acceptability of bupropion/naltrexone in this population and potential efficacy signals.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 21 and 34 years.
2. A minimum of 5/3 (men/women) or more binge drinking episodes per month over the past three months. A binge drinking episode is defined as the consumption of 5/4 (men/women) standard drinks (~12 gms ethanol) in about a two hour period. Subjects may meet DSM-V criteria for mild or moderate alcohol use disorder.
3. Ability to understand and sign written informed consent.
4. Must have a 0.0 gms/dl breathalyzer reading on the day of screening and 0.0 gms/dl on the day of randomization.
5. Must have a stable residence and be able to identify an individual who could contact participant if needed.
6. Have a goal of sobriety or significantly reducing alcohol intake.

Exclusion Criteria

1. Presence of physical dependence on alcohol as assessed by clear tolerance to alcohol or alcohol withdrawal symptoms based on SCID interview or a Severe Alcohol Use Disorder (>5 SCID DSM-V symptoms).
2. Bupropion is contraindicated in individuals with a history of bulimia or a seizure disorder and naltrexone is contraindicated in acute liver disease and in patients using or misusing opioids.
3. Clinically significant medical disease that might interfere with the evaluation of the study medication or present a safety concern (e.g., renal insufficiency, cirrhosis, unstable hypertension, diabetes mellitus, seizure disorder). Clinically significant psychiatric illness including any psychotic disorder, bipolar disorder, anorexia/bulimia, severe depression, or suicidal ideation.
4. Other substance abuse or dependence disorder other than nicotine or cannabis abuse.
5. Concurrent use of anticonvulsants. Concurrent use of any psychotropic medication including antidepressants, mood stabilizers, antipsychotics, anxiolytics, stimulants, or hypnotics with the exception of stable doses of antidepressants for one month. Bupropion is commonly added to antidepressants for augmentation so the use of another antidepressant does not represent a safety concern. Prior history of adverse reaction to bupropion or naltrexone.
6. AST or ALT > 3.5 times ULN or bilirubin > 1.5 X ULN.
7. Positive urine toxicology screen with the exception of cannabis. Individuals with positive cannabis screens will be excluded only if they have a history of cannabis dependence.
8. Pregnant women and women of childbearing potential who do not practice a medically acceptable form of birth control (oral or depot contraceptive, or barrier methods such as diaphragm or condom with spermicidal).
9. Women who are breastfeeding.
10. Individuals requiring inpatient treatment or more intense outpatient treatment for their alcohol problems.
11. Participation in any clinical trial within the past 60 days that would have safety concerns for the trial.
12. Court-mandated participation in alcohol treatment or pending incarceration.

Ages: 21 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Garbutt, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Naltrexone and Buproprion: Bupropion XL 150 mg/d on Days 1-4 increased to 300 mg/d for Days 5-84. Naltrexone 25 mg/d from Days 7-9 and increased to 50 mg/d for Days 10-84.
Period: Overall Study
Arm/Group | Naltrexone and Buproprion
Started | 12
Completed | 11
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Naltrexone and Buproprion
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
Number of Binge Drinking Days in 90 days prior to screening [Mean (Standard Deviation); unit: days] | 17.3 (7.8)
Intensity of Binge Drinking prior to Study [Mean (Standard Deviation); unit: drinks/binge drinking day] — The mean number of drinks/binge drinking day in the 90 days prior to screening.
  drinks/binge drinking day | 8.4 (1.0)
Craving for Alcohol [Mean (Standard Deviation); unit: units on a scale] — The PACS is a five-item self-administered instrument for assessing craving. Frequency, intensity, and duration of thoughts about drinking are assessed along with ability to resist drinking. The final item asks the responder to provide an average rating of his/her craving over the course of the past week. The questions on the PACS use descriptors coupled with numerical ratings ranging from 0 to 6 with the highest possible total score of 30. Higher scores reflect a higher level of craving.
  units on a scale | 11.25 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Associated Adverse Events
Description: Tolerability assessed by specifically probing for intervention-associated adverse effects.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Naltrexone and Buproprion
Number analyzed (Participants) | 12
Participants
  Headache | 5
  Insomnia | 2
  Dizziness | 2

2. Primary Outcome: Number of Participants Discontinuing Subsequent to Defined Intolerance
Description: Retention was evaluated indirectly by accounting for those participants who discontinued either naltrexone or bupropion or study participation itself due to intolerance.
Time Frame: Throughout study, a total of approximately 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Naltrexone and Buproprion
Number analyzed (Participants) | 12
Participants
  Discontinued: Naltrexone | 3
  Discontinued: Buproprion | 1
  Discontinued: Study | 1

3. Primary Outcome: Number of Binge Drinking Days During Treatment
Description: The number of binge drinking days during treatment with bupropion + naltrexone
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Naltrexone and Buproprion
Number analyzed (Participants) | 12
days | 3.2 (2.9)

4. Secondary Outcome: Final Penn Alcohol Craving Scale (PACS) Score
Description: Craving for alcohol will be assessed using the Penn Alcohol Craving Scale (PACS) The PACS is a five-item self-administered instrument for assessing craving. Frequency, intensity, and duration of thoughts about drinking are assessed along with ability to resist drinking. The final item asks the responder to provide an average rating of his/her craving over the course of the past week. The questions on the PACS use descriptors coupled with numerical ratings ranging from 0 to 6 with the highest possible total score of 30. Higher scores reflect a higher level of craving. This outcome measure is the final PACS total score obtained in the trial.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naltrexone and Buproprion
Number analyzed (Participants) | 12
units on a scale | 4.4 (4.2)

5. Secondary Outcome: Mean Number of Drinks/Binge Drinking Day During Treatment
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: drinks/binge drinking day
Arm/Group | Naltrexone and Buproprion
Number analyzed (Participants) | 12
drinks/binge drinking day | 3.3 (0.9)

ADVERSE EVENTS:
Time Frame: Throughout the 12-week study period.
Arm/Group | Naltrexone and Buproprion
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 11/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone and Buproprion (N=12)
Headache (Nervous system disorders) | 5 (5)
Insomnia (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Low energy (General disorders) | 2 (2)
Reduced Appetite (General disorders) | 1 (1)
Dry Mouth (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Irritability (Nervous system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT02842073/Prot_SAP_000.pdf